CLINICAL TRIAL: NCT04280341
Title: A Phase I, Open-label, Dose Escalation Clinical Trial to Assess the Safety, Efficacy, Tolerability and Pharmacokinetics of the Recombinant Humanized Anti-PD1 Monoclonal Antiody (JS001) in Combination With Recombinant Humanized Anti-HER2 Monoclonal Antibody-MMAE Conjugate (RC48-ADC) in Treatment of HER2-Positive Advanced Malignant Solid Tumors
Brief Title: JS001 in Combination With RC48-ADC in Treatment of HER2-Positive Advanced Malignant Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University (Other)
Collaborators: RemeGen Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Shen Lin, MD，Professor,Chief of Department of GI Oncology,Peking University Cancer Hospital, Peking University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RC48-C013
Record Dates: First submitted 2019-12-30; First posted 2020-02-21 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: HER2-Positive Solid Tumors
Keywords: RC48-ADC; JS001; HER2 positive solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RC48-ADC in combinaton with Anti-PD1 Monoclonal Antibody (Experimental): RC48-ADC(Recombinant Humanized Anti-HER2 Monoclonal Antibody-MMAE Conjugate) JS001(Recombinant Humanized Anti-PD1 Monoclonal Antibody)
  Interventions: Biological: RC48-ADC in combinaton with JS001

INTERVENTIONS:
Biological: RC48-ADC in combinaton with JS001 — The study has 2 parts which include dose escalation phase and dose extension phase.
  Dose escalation will use a 3+3 design and will enroll cohorts of 3-6 patients with HER2-Positive Advanced Malignant Solid Tumors sequentially at escalating doses of 2.0mg/kg and 2.5mg/kg to RC48-ADC and JS001 is fixed dose of 3.0mg/mg

SUMMARY:
This is a non-randomized, open-label, single-arm, multicenter Phase I clinical trial which will evaluate the Safety, Efficacy, Tolerability and Pharmacokinetics of RC48-ADC in combinaton with Anti-PD1 Monoclonal Antibody in Treatment of HER2-Positive Advanced Malignant Solid Tumors.

DETAILED DESCRIPTION:
The study has 2 parts which include dose escalation phase and dose extension phase.

Dose escalation will use a 3+3 design and will enroll cohorts of 3-6 patients with HER2-Positive Advanced Malignant Solid Tumors sequentially at escalating doses of 2.0mg/kg and 2.5mg/kg to RC48-ADC and JS001 is fixed dose of 3.0mg/mg . Escalation will continue until identification of a MTD.

Dose of phase II and extenstion stage which based-results of escalation phase will be recommend.

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign the informed consent form;
* ≥18 years old;
* Diagnosed histologically or cytologically with local advanced or metastatic HER2-positive malignant solid cancer( indicating that IHC result is 2+,3+or1+ ) and under one of following situations: standard treatment-refractory (disease progression or no response), treatment-resistant, unable to receive treatment, or the standard treatment is unavailable;
* Having measurable or evaluable lesions according to RECIST 1.1;
* Having an ECOG performance status score of 0 or 1;
* Echocardiographic LVEF (left ventricular ejection fraction) ≥ 50%.
* NYHA CLAS 0-1;
* Having sufficient bone marrow, liver and kidney functions (based on the normal value of the clinical trial site) within 7 days before erollment: Absolute neutrophil count (ANC) ≥ 1.5×109/L,Platelets ≥ 100×109/L, hemoglobin≥ 9.0 g/dL；Total serum bilirubin ≤ 1.5×upper limit of normal (ULN);Without liver metastasis, ALT, AST or ALP ≤ 2.5×ULN; With liver metastasis, ALT, AST or ALP ≤ 5×ULN;Serum creatinine clearance rate ≥ 60 mL/min(Cockcroft-Gault formula);INR International Normalized Ratio ≤ 1.5 × ULN, APTT ≤ 1.5 × ULN;
* With an expected survival of more than 3 months;
* Male or female patients of childbearing potential must agree to use effective methods of contraception (such as double-barrier contraceptive methods, condoms, oral or injectable contraceptives and intrauterine devices) during the study period and within 24 weeks after the last dosing;

Exclusion Criteria:

* Known active uncontrolled or symptomatic CNS metastases, as indicated by clinical symptoms, cerebral edema, spinal cord compression, carcinomatous meningitis, leptomeningeal disease and/or progressive growth. Patients with a history of CNS metastases or cord compression are eligible if they have been definitively treated and are clinically stable o before the first dose of RC48-ADC.
* Prior treatment with HER2 targeted therapy while LVEF decline <45% or absolute value of LVEF decline >15%；
* Participation in any other studies within 4 weeks before study entry and/or during participation in the active treatment phase of the trial.
* Radical operation within 3 weeks before study entry but not include diagnostic puncture or peripheral vascular assess replacement ;
* Radical radiation therapy within 3 months before study entry; Patient of Palliative radiotherapy is eligible into this study if <30 % Radiation area of bone marrow;
* Patients who underwent checkpoint inhibitor or tumor vaccines include not limited PD-1、 PD-1、PD-L1、CTLA4、LAG3;
* Patient has had systemic steroid therapy (≥10 mg/day of prednisone or physiologic replacement doses of hydrocortisone, or its equivalent) or immunosuppressive medication within 14 days prior to the first dose of study.
* Live vaccines within 28 days prior to the first dose of study and during trial treatment.
* Patient has an active autoimmune disease or a documented history of autoimmune disease (but not limited In terstitial lung Disease, uveitis, SLE, etal). Patients with vitiligo or resolved childhood asthma/atopy would be exception to this rule. Patients that require inhaled steroids or local steroid injections would not be excluded from the study. Patients with vitiligo or psoriasis that is stable on hormone replacement will not be excluded from the study.
* Active and clinically significant bacterial, fungal or viral infection including hepatitis B (HBV), hepatitis C (HCV), known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS)-related illness.
* Patients have uncontrollable systemic disease which including diabetes, hypertendion, pulmonary fibrosis, etal.
* The toxicity of previous anti-cancer therapy has not returned to 0 or 1 level as specified in CTCAE v4.0 (except for hair loss);
* Patient has a history of allogeneic HSCT or organ transplation before study entry;
* Patients with hypersensitivity or delayed hypersensitivity reactions to certain components of RC48-ADC or similar drugs;
* Patients with symptomatic include but not limited ascites or pleural effusion and mental disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-06-03 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
DLT(dose-limiting toxicity) or Maximal Tolerance Dose (MTD) | 28 days
  Side effects of drug or treatment that are serious enough to prevent an increase in dose or level of that treatment. The MTD is defined as the previous dose level.
adverse events | 1 year
  Safety of participants followed for the duration of hospital stay, an expected average of 1 week

SECONDARY OUTCOMES:
ORR | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  Percentage of patients who achieve partial response (PR) or complete response (CR) based on Response Evaluation Criteria In Solid Tumors (RECIST v1.1).
DOR | From date of first dose until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  The percentage of patients who achieve complete remission(CR) or partial remission
PFS | up to 2 years
  progression free survival
OS | up to 2 years
  overall survival
ADA | up to 2 years
  anti-drug antibody which can result in treatment failure by blocking the pharmacological function of the drug.
NADA | up to 2 years
  neutralizing anti-drug antibody which can result in treatment failure by blocking the pharmacological function of the drug.
Cmax | up to 3 cycles(each cycle is 14 days)
  Peak plasma concentration
AUC | up to 3 cycles(each cycle is 14 days)
  area under the plasma concentration versus time curve
Tmax | up to 3 cycles(each cycle is 14 days)
  Time for peak concentration

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, professor, Principal Investigator — Peking University
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Wang Y, Gong J, Wang A, Wei J, Peng Z, Wang X, Zhou J, Qi C, Liu D, Li J, Lu M, Lu Z, Cao Y, Yuan J, Zhang R, Fang J, Zhang X, Shen L. Disitamab vedotin (RC48) plus toripalimab for HER2-expressing advanced gastric or gastroesophageal junction and other solid tumours: a multicentre, open label, dose escalation and expansion phase 1 trial. EClinicalMedicine. 2024 Jan 5;68:102415. doi: 10.1016/j.eclinm.2023.102415. eCollection 2024 Feb. PMID 38235421